CLINICAL TRIAL: NCT02293356
Title: Phase IV Clinical Trial of Nimotuzumab in the Treatment of Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-Nim-NPC-2
Record Dates: First submitted 2014-10-31; First posted 2014-11-18 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab Injection (Experimental): 200mg,Once a week，Intravenous infusion over 60 minutes
  Interventions: Drug: Nimotuzumab Injection

INTERVENTIONS:
Drug: Nimotuzumab Injection — patients receive nimotuzumab injection for 200mg/w,intravenous infusion over 60 minutes.Doctor adjust the dosage of nimotuzumab and choose other treatment options according to the actual situation of patients.
  Other Names: Taixinsheng

SUMMARY:
This clinical study is designed as an open, single group, multi-center, phase 4 clinical study to assess the safety of Nimotuzumab in the treatment of nasopharyngeal carcinoma and to provide a more reasonable basis for clinical drug programs.

DETAILED DESCRIPTION:
This clinical study is designed as an open, single group, multi-center, phase 4 clinical study to assess the safety of Nimotuzumab in the treatment of nasopharyngeal carcinoma and to provide a more reasonable basis for clinical drug programs.

Subjects who meet the inclusion/exclusion criteria are administered of Nimotuzumab based on medication instructions or adjusted by clinicians according to the treatment. In case of the progression of disease, unacceptable toxicity, withdrawal of the consent, or judgment by investigator that the treatment needs to be stopped, the treatment of Nimotuzumab is stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed nasopharyngeal carcinoma
2. Sex and age without limiting
3. Treatment without limiting
4. Subjects with reproductive potential (males and females) willing to use reliable means of contraception
5. Able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

1. Patients with severe allergies or idiosyncratic constitution
2. Women who are pregnant (determined by urine pregnancy test)or breast feeding
3. Any other severe complications or functional disorder of organ systems, which will affect the evaluation of safety of patients or will interfere with the test drug according to the researcher's point of view

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of the treatment with Nimotuzumab(NCI Common Terminology Criteria for Adverse Events v4.03) | up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: li gao, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute & Hospital.Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China